CLINICAL TRIAL: NCT03075410
Title: A Double Blind, Placebo-controlled First Time in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of GSK3036656 in Healthy Adult Volunteers
Brief Title: First Time in Human (FTIH) Safety and Pharmacokinetics (PK) Study of GSK3036656 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 201040; 2015-003654-41 (EudraCT Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Tuberculosis
Keywords: ascending dose; Pharmacokinetics; GSK3036656; FTIH; Safety
MeSH Terms: conditions — Tuberculosis | interventions — GSK656

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Cohort 1- GSK3036656 in Part A (Experimental): During Part A (Cohort 1), Subjects will receive a single dose of GSK3036656 in the morning on Day 1 in each of the 4 treatment (dosing) periods after an overnight fast of at least 8 hours. Dosing with food may also be done in Part A once results from the food effect analysis are available. The total daily dose for the treatment (dosing) period may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. The starting dose in Part A will be 5 mg and will then be escalated up to a dose no higher than 1500 mg. One of the 4 dosing periods will be food effect group which will be determined based on from previous cohorts. For the food effect assessment, the selected dose will be given with a high fat meal. There will be a 2 week washout between doses initially but the washout period may be modified depending on emerging data from previous cohorts. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 1- Placebo in Part A (Placebo Comparator): During Part A (Cohort 1), Subjects will receive a single matching placebo in morning on Day 1 in each of the 4 treatment (dosing) periods after an overnight fast of at least 8 hours. Dosing with food may also be done in Part A once results from the food effect analysis are available. Placebo for the treatment (dosing) period may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same period. One of the 4 dosing periods will be food effect group which will be determined based on from previous cohorts. For the food effect assessment, placebo will be given with a high fat meal. There will be a 2 week washout between doses initially but the washout period may be modified depending on emerging data from previous cohorts. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo
- Cohort 2- GSK3036656 in Part A (Experimental): During Part A (Cohort 2), Subjects will receive a single dose of GSK3036656 in morning on Day 1 in each period after an overnight fast of at least 8 hours. Dosing with food may also be done once results from the food effect analysis are available. The total dose for the treatment period may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. The dose will be selected on basis of safety, tolerability and PK data from the previous treatment period or cohort and will then be escalated up to a dose no higher than 1500 mg. One of the 4 dosing periods will be food effect group, determined based on from previous cohorts, where the selected dose will be given with a high fat meal. There will be a 2 week washout between doses initially but the washout period may be modified depending on emerging data from previous cohorts. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 2- Placebo in Part A (Placebo Comparator): During Part A (Cohort 2), Subjects will receive a single matching placebo in morning on Day 1 in each of the 4 treatment (dosing) periods after an overnight fast of at least 8 hours. Dosing with food may also be done once results from the food effect analysis are available. Placebo for the treatment period may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same period. One of the 4 dosing periods will be food effect group, determined based on from previous cohorts, where the placebo will be given with a high fat meal. There will be a 2 week washout between doses initially but the washout period may be modified depending on emerging data from previous cohorts. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo
- Cohort 3- GSK3036656 in Part B (Experimental): During Part B (Cohort 3), Subjects will receive a single dose of GSK3036656 once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive repeat single dose of GSK3036656 once daily over a period of 14 days. Dosing with food may also be done if there are PK or tolerability reasons making it preferable to dose in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. Appropriate dose and dose regimen will be selected on available safety, tolerability and PK data from Part A. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 3- Placebo in Part B (Placebo Comparator): During Part B (Cohort 3), Subjects will receive a single matching placebo once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive a placebo once daily over a period of 14 days. Dosing with food may also be done if the active treatment is given in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same cohort. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo
- Cohort 4- GSK3036656 in Part B (Experimental): During Part B (Cohort 4), Subjects will receive a single dose of GSK3036656 once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive repeat single dose of GSK3036656 once daily over a period of 14 days. Dosing with food may also be done if there are PK or tolerability reasons making it preferable to dose in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. Appropriate dose and dose regimen will be selected on available safety, tolerability and PK data from preceding repeat dose cohorts from Part B. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 4- Placebo in Part B (Placebo Comparator): During Part B (Cohort 4), Subjects will receive a single matching placebo once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive a placebo once daily over a period of 14 days. Dosing with food may also be done if the active treatment is given in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same cohort. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo
- Cohort 5- GSK3036656 in Part B (Experimental): During Part B (Cohort 5), Subjects will receive a single dose of GSK3036656 once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive repeat single dose of GSK3036656 once daily over a period of 14 days. Dosing with food may also be done if there are PK or tolerability reasons making it preferable to dose in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. Appropriate dose and dose regimen will be selected on available safety, tolerability and PK data from preceding repeat dose cohorts from Part B. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 5- Placebo in Part B (Placebo Comparator): During Part B (Cohort 5), Subjects will receive a single matching placebo once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive a placebo once daily over a period of 14 days. Dosing with food may also be done if the active treatment is given in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same cohort. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo
- Cohort 6- GSK3036656 in Part B (Experimental): During Part B (Cohort 6), Subjects will receive a single dose of GSK3036656 once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive repeat single dose of GSK3036656 once daily over a period of 14 days. Dosing with food may also be done if there are PK or tolerability reasons making it preferable to dose in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours on discretion of the GSK study team and the principal investigator. Appropriate dose and dose regimen will be selected on available safety, tolerability and PK data from preceding repeat dose cohorts from Part B. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: GSK3036656
- Cohort 6- Placebo in Part B (Placebo Comparator): During Part B (Cohort 6), Subjects will receive a single matching placebo once daily in morning on Day 1 after an overnight fast of at least 8 hours. Subjects will receive a placebo once daily over a period of 14 days. Dosing with food may also be done if the active treatment is given in a fed state (dose will be given with a high fat meal.). The total dose may also be divided into 2 or 3 smaller doses administered within 24 hours in a similar manner if divided for subjects receiving active treatment in the same cohort. Subjects will be followed up to 2 weeks from the last dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3036656 — GSK3036656 is available as capsules (for oral administration) containing 5 mg, 25 mg or 100 mg of GSK3036656 as free base equivalent.
  Arms: Cohort 1- GSK3036656 in Part A; Cohort 2- GSK3036656 in Part A; Cohort 3- GSK3036656 in Part B; Cohort 4- GSK3036656 in Part B; Cohort 5- GSK3036656 in Part B; Cohort 6- GSK3036656 in Part B
Drug: Placebo — Placebo is a matching capsule containing Avicel PH (Suitable for Pharmaceutical Use) 102, for oral administration.
  Arms: Cohort 1- Placebo in Part A; Cohort 2- Placebo in Part A; Cohort 3- Placebo in Part B; Cohort 4- Placebo in Part B; Cohort 5- Placebo in Part B; Cohort 6- Placebo in Part B

SUMMARY:
GSK3036656 is being developed by GSK for the treatment of tuberculosis (TB). This is the FTIH study for GSK3036656 to evaluate the safety, tolerability and PK of single ascending and repeat oral doses of GSK3036656 in healthy adult subjects. The results of this study are intended to be used to identify appropriate and well-tolerated doses of GSK3036656 to be used in further studies. A food effect assessment will also be undertaken to investigate the influence of food on the PK of GSK3036656. The study will be conducted in two parts: Part A (single dose) and Part B (repeat dose). Up to two cohorts will be included in Part A. 9 healthy adult subjects will be included in each cohort. Each cohort will participate in up to 4 treatment (dosing) periods including a food effect treatment period. During each treatment period, GSK3036656 will be administered to 6 subjects and placebo will be administered to 3 subjects. The starting dose in Part A will be 5 milligrams (mg), and the maximum dose will be 1500 mg. The two cohorts in Part A will be dosed sequentially (i.e., dosing in Cohort 2 starts after dosing in Cohort 1 is completed). Initially, there will be a 14 day wash out period for individual subjects between each dose level. Study progression to Part B from Part A will be based on an acceptable safety, tolerability and PK profile in Part A. Part B will comprise up to 4 cohorts (Cohorts 3, 4, 5, and 6) each containing 10 (8 active: 2 placebo) healthy adult subjects to examine the safety, tolerability and PK of a repeated daily dose of GSK3036656 over a period of up to 14 days. Appropriate doses and dose regimens for Part B will be selected based on available safety, tolerability and PK data from Part A and/or any preceding repeat dose cohorts from Part B. Dividing the total daily dose into 2 or 3 smaller doses may be done in both Part A and Part B. Up to 18 subjects will be enrolled into Part A and up to 40 subjects will be enrolled into Part B. The total duration of the study for each subject recruited into Part A and Part B will be approximately 12 weeks and 8 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied, may be included only if the investigator in consultation with the medical monitor, if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=60 kilograms (kg) and body mass index (BMI) within the range 19 to 29.9 kg/meter^2 inclusive.
* Male
* Female subjects of non-child bearing potential are eligible to participate. Non-child bearing potential is defined as:

  * Pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or documented bilateral salpingectomy; hysterectomy; documented bilateral oophorectomy.
  * Postmenopausal defined as 12 months of spontaneous amenorrhea. Post-menopausal status will be confirmed by a simultaneous follicle stimulating hormone (FSH) and estradiol levels test.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 90 days after the last dose of study treatment (i.e. one sperm cycle).

  * Vasectomy with documentation of azoospermia.
  * Male condom plus partner use of one of the contraceptive options as follows: contraceptive subdermal implant; intrauterine device or intrauterine system; highly effective oral contraceptive, either combined or progestogen alone (provided it is associated with inhibition of ovulation); injectable progestogen; contraceptive vaginal ring; percutaneous contraceptive patches.
* These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5 times of upper limit of normal (ULN) (isolated bilirubin >1.5 times of ULN may be acceptable, after consultation with the GlaxoSmithKline (GSK) medical monitor, if bilirubin is fractionated and direct bilirubin <35 percent)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF >450 milliseconds.
* Presence of moderate or severe valve disorder or any other clinically significant abnormality.
* Subjects with a history of photosensitivity.
* Females of non-childbearing potential who are susceptible to heavy periods or vaginal bleeding or spotting.
* Pregnant females. A human chorionic gonadotrophin (hCG) test will be performed on Day -1 of each treatment (dosing) period in Part A and Part B for women for whom post-menopausal status has not been confirmed by FSH/estradiol testing. No pregnancy tests will be required for female subjects confirmed as post-menopausal by FSH/estradiol testing.
* Lactating females.
* Use of prescription or non-prescription drugs, including high-dose vitamins, herbal and dietary supplements (including Saint John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and sponsor, the medication will not interfere with the study procedures or compromise subject safety. Paracetamol for mild analgesia will be permitted.
* Breath carbon monoxide test indicative of smoking or history of current use of tobacco- or nicotine-containing products.
* Current regular alcohol consumption defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Subjects must not sunbathe or use a tanning device whilst taking the study medication and until at least 2 weeks after their last dose. Subjects are to be advised that they should wear protective clothing (e.g. sun hat, long sleeves) and use a broad spectrum ultraviolet A/ ultraviolet B sunscreen (sun protection factor >=30) when outdoors.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive test for human immunodeficiency virus (HIV) antibody.
* A positive pre-study drug/alcohol screen.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Tenero D, Derimanov G, Carlton A, Tonkyn J, Davies M, Cozens S, Gresham S, Gaudion A, Puri A, Muliaditan M, Rullas-Trincado J, Mendoza-Losana A, Skingsley A, Barros-Aguirre D. First-Time-in-Human Study and Prediction of Early Bactericidal Activity for GSK3036656, a Potent Leucyl-tRNA Synthetase Inhibitor for Tuberculosis Treatment. Antimicrob Agents Chemother. 2019 Jul 25;63(8):e00240-19. doi: 10.1128/AAC.00240-19. Print 2019 Aug. PMID 31182528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double blind, placebo-controlled study to evaluate the safety, tolerability and pharmacokinetics (PK) of single and repeat doses of GSK3036656 in healthy adult participants. The study was conducted at 1 center in United Kingdom from 02-April-2017 to 04-August-2017. Part A was a crossover design, Part B was a parallel group design..
Pre-assignment Details: 20 participants screened, 8 were screen failures (SF). 9 were randomized at the beginning of Part A. During Part A, 2 of the 3 participants who withdrew were replaced, hence 11 randomized. 30 participants screened, 7 were SF, 4 passed screening but were kept in reserve, hence 19 randomized in Part B.
Groups:
- PartA - Placebo/15 mg/25 mg/5 mg (Fed): Participants received matching placebo to GSK3036656 5 milligrams (mg) followed by GSK3036656 15 mg followed by GSK3036656 25 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- PartA - Placebo/15 mg/25 mg/Placebo: Participants received matching placebo to GSK3036656 5 mg followed by GSK3036656 15 mg followed by GSK3036656 25 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- PartA - 5 mg/Placebo/25 mg/5 mg (Fed): Participants received SK3036656 5 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 25 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- PartA - 5 mg/Placebo/25 mg/Placebo: Participants received SK3036656 5 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 25 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- PartA - 5 mg/15 mg/Placebo/5 mg (Fed): Participants received GSK3036656 5 mg followed by GSK3036656 15 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- PartA - 5 mg/15 mg/Placebo/Placebo: Participants received GSK3036656 5 mg followed by GSK3036656 15 mg followed by matching placebo to GSK3036656 5 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- Part B-Placebo: Participants received matching placebo to active GSK3036656 5 mg / 15mg capsules orally once daily for 14 days.
- Part B-Repeat GSK3036656 5 mg: Participants received repeat dosing of GSK3036656 5 mg capsules orally once daily for 14 days.
- Part B-Repeat GSK3036656 15 mg: Participants received repeat dosing of GSK3036656 15 mg capsules orally once daily for 14 days.
Period: Part A-Period 1 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Washout Period 1 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Period 2 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Personal reasons | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Washout Period 2 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Period 3 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 2 (Participants who withdrew in Period 2 were replaced (2 new participants entered Part A period 3).) | 1 | 2 (Participants who withdrew in Period 2 were replaced (2 new participants entered Part A period 3).) | 1 | 2 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reaction to ECG tabs causing a rash | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Washout Period 3 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A-Period 4 (14 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (up to 28 Days)
Arm/Group | PartA - Placebo/15 mg/25 mg/5 mg (Fed) | PartA - Placebo/15 mg/25 mg/Placebo | PartA - 5 mg/Placebo/25 mg/5 mg (Fed) | PartA - 5 mg/Placebo/25 mg/Placebo | PartA - 5 mg/15 mg/Placebo/5 mg (Fed) | PartA - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 9 participants were randomized at the beginning of Part A. During Part A, 2 of the 3 participants who withdrew were replaced, hence 11 randomized.
Groups:
- Part A - Placebo/15 mg/25 mg/5 mg (Fed): Participants received matching placebo to GSK3036656 5 mg followed by GSK3036656 15 mg followed by GSK3036656 25 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- Part A - Placebo/15 mg/25 mg/Placebo: Participants received matching placebo to GSK3036656 5 mg followed by GSK3036656 15 mg followed by GSK3036656 25 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- Part A - 5 mg/Placebo/25 mg/5 mg (Fed): Participants received SK3036656 5 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 25 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- Part A - 5 mg/Placebo/25 mg/Placebo: Participants received SK3036656 5 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 25 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- Part A - 5 mg/15 mg/Placebo/5 mg (Fed): Participants received GSK3036656 5 mg followed by GSK3036656 15 mg followed by matching placebo to GSK3036656 5 mg followed by GSK3036656 5 mg (fed) capsules orally for 14 Days.
- Part A - 5 mg/15 mg/Placebo/Placebo: Participants received GSK3036656 5 mg followed by GSK3036656 15 mg followed by matching placebo to GSK3036656 5 mg followed by matching placebo to GSK3036656 5 mg capsules orally for 14 Days.
- Total: Total of all reporting groups
Arm/Group | Part A - Placebo/15 mg/25 mg/5 mg (Fed) | Part A - Placebo/15 mg/25 mg/Placebo | Part A - 5 mg/Placebo/25 mg/5 mg (Fed) | Part A - 5 mg/Placebo/25 mg/Placebo | Part A - 5 mg/15 mg/Placebo/5 mg (Fed) | Part A - 5 mg/15 mg/Placebo/Placebo | Part B-Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg | Total
Number analyzed (Participants) | 3 | 1 | 3 | 1 | 2 | 1 | 4 | 7 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (5.03) | 25 (NA) — Standard deviation was not calculated as a single participant was analyzed. | 26.3 (2.52) | 28.0 (NA) — Standard deviation was not calculated as a single participant was analyzed. | 34.0 (1.41) | 50.0 (NA) — Standard deviation was not calculated as a single participant was analyzed. | 30.3 (9.43) | 31.9 (6.26) | 35.1 (7.88) | 32.5 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Male | 3 | 1 | 3 | 1 | 2 | 0 | 4 | 7 | 8 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian-South Asian Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Black/ African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White-White/Caucasian/European Heritage | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 5 | 8 | 23
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (nSAE) and Serious Adverse Events (SAEs) for Part A
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above. Safety Population comprised of all randomized participants who received at least one dose of study medication.
Time Frame: Up to 12 weeks
Population: Safety Population for Part A
Measure: Count of Participants; unit: Participants
Groups:
- Part A-Matching Placebo: Participants received single dosing of matching placebo to GSK3036656 5 mg capsules orally.
- Part A-GSK3036656 5 mg: Participants received single dosing of GSK3036656 5 mg capsules orally.
- Part A-GSK3036656 15 mg: Participants received single dosing of GSK3036656 15 mg capsules orally.
- Part A-GSK3036656 25 mg: Participants received single dosing of GSK3036656 25 mg capsules orally.
- Part A-GSK3036656 5 mg (Fed): Participants received single dosing of GSK3036656 5 mg capsules in the fed state orally.
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants
  nSAE | 1 | 1 | 1 | 3 | 1
  SAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With nSAE and SAEs for Part B
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above.
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Groups:
- Part B-Matching Placebo: Participants received matching placebo to active GSK3036656 5 mg / 15mg capsules orally once daily for 14 days.
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  nSAE | 0 | 2 | 1
  SAE | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings for Part A
Description: 12-lead ECGs were collected during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) intervals. At each time point at which triplicate ECGs were required, three individual ECG tracings were obtained as closely as possible in succession, but no more than 2 to 5 minutes apart. ECG findings were categorized as normal, abnormal not clinically significant (A-NCS) and abnormal clinically significant (A-CS). Only A-NCS and A-CS worst case post-Baseline values have been presented. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Up to 6 weeks
Population: Safety Population for Part A. For arm Part A-Matching Placebo 3 of the 9 placebo participants received placebo twice, therefore they had these measures done in 2 different treatment periods, so N=9 but number of units analyzed=12.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants
  A-NCS | 2 | 1 | 0 | 0 | 0
  A-CS | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects With Clinically Relevant Changes in ECG in Part B
Description: 12-lead ECGs were collected during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT interval and QTcF intervals. At each time point at which triplicate ECGs were required, three individual ECG tracings were obtained as closely as possible in succession, but no more than 2 to 5 minutes apart. ECG findings were categorized as normal, A-NCS and A-CS. Only A-NCS and A-CS worst case post-Baseline values have been presented.
Time Frame: Up to 8 weeks
Population: Safety Population for Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  A-NCS | 1 | 3 | 3
  A-CS | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Cardiac Telemetry Findings for Part A
Description: Continuous cardiac telemetry was performed from approximately 1 hour pre-dose to 24 hours post dosing . Number of participants who had abnormal findings upon cardiac telemetry assessment have been presented.
Time Frame: 25 hours for each period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Cardiac Telemetry Findings for Part B
Description: as for outcome 5
Time Frame: 25 hours for each period
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Vital Sign Parameters Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) of Potential Clinical Importance (PCI) for Part A
Description: SBP and DBP were assessed in supine position with a completely automated device. Measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones). The PCI range for SBP was less than 85 mmHg (lower) and greater than 160 mmHg (upper) while that for DBP was less than 45 mmHg (lower) and greater than 100 mmHg (upper).
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants
  SBP | 0 | 0 | 0 | 0 | 0
  DBP | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Vital Sign Parameters SBP and DBP of PCI for Part B
Description: as for outcome 7
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  SBP | 0 | 0 | 0
  DBP | 0 | 0 | 1

9. Primary Outcome: Number of Participants With Vital Sign Parameter Heart Rate of PCI for Part A
Description: Heart rate was assessed in supine position with a completely automated device. Measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones). The PCI range for heart was less than 40 bpm (lower) and greater than 110 bpm (upper).
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Vital Sign Parameter Heart Rate of PCI for Part B
Description: as for outcome 9
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Vital Sign Parameter Temperature of PCI for Part A
Description: Number of participants with temperature data of PCI have been presented.
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Vital Sign Parameter Temperature of PCI for Part B
Description: Number of participants with temperature data of PCI have been presented.
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of PCI for Part A
Description: Blood samples were collected for the assessment of clinical chemistry parameters namely blood urea nitrogen (BUN), creatinine, glucose, cholesterol, potassium, sodium, calcium, aspartate amino transferase (AST), alanine amino transferase (ALT), alkaline phosphatase, triglycerides, total and direct bilirubin, total protein, albumin and troponin. Only categories with PCI values have been presented, therefore only AST is presented.
Time Frame: Up to 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 1

14. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of PCI for Part B
Description: Blood samples were collected for the assessment of clinical chemistry parameters namely BUN, creatinine, glucose, cholesterol, potassium, sodium, calcium, AST, ALT, alkaline phosphatase, triglycerides, total and direct bilirubin, total protein, albumin and troponin. Only categories with PCI values have been presented.
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  ALT | 0 | 1 | 0
  AST | 0 | 1 | 0

15. Primary Outcome: Number of Participants With Hematology Parameters of PCI for Part A
Description: Blood samples were collected for the assessment of hematology parameters platelet count, red blood cell count, hemoglobin, hematocrit, reticulocytes, mean corpuscle volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, basophils and eosinophils. Only categories with PCI values have been presented.
Time Frame: Up to 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Hematology Parameters of PCI for Part B
Description: as for outcome 15
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  Leukocytes | 0 | 1 | 0
  Neutrophils | 0 | 1 | 1

17. Primary Outcome: Number of Participants With Abnormal Urinalysis Parameters for Part A
Description: Urinalysis included dipstick urine test which was used to screen for glucose, ketones, occult blood and protein up to 72 hours post dose. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose, ketones, occult blood and protein can be read as negative, trace, trace-intact, trace-lysed,1+ and 2+ indicating proportional concentrations in the urine sample. Only categories with non-negative values have been presented. Only those participants with data available the indicated time points were analyzed.
Time Frame: Up to 72 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
Participants
  Day -1, Ketone, Trace | 1 | 0 | 1 | 0 | 0
  Day -1, Occult blood, 1+ | 0 | 0 | 0 | 0 | 1
  Day -1, Occult blood, 2+ | 0 | 0 | 1 | 0 | 0
  Day -1, Occult blood, trace-intact | 1 | 0 | 0 | 0 | 0
  Day -1, Occult blood, trace-lysed | 1 | 0 | 0 | 0 | 0
  Day -1, Protein, Trace | 1 | 0 | 2 | 0 | 1
  24 hours, Ketones, 2+ | 1 | 0 | 0 | 0 | 0
  24 hours, Occult blood, 2+ | 0 | 0 | 1 | 0 | 0
  24 hours, Occult blood, trace-intact | 1 | 0 | 0 | 0 | 0
  24 hours, Occult blood, trace-lysed | 1 | 0 | 0 | 0 | 0
  72 hours, Ketone, Trace | 0 | 0 | 1 | 0 | 0
  72 hours, Occult blood, 1+ | 1 | 0 | 1 | 0 | 0
  72 hours, Occult blood, trace-intact | 0 | 0 | 0 | 0 | 1
  72 hours, Occult blood, trace-lysed | 0 | 0 | 0 | 1 | 0
  72 hours, Protein, Trace | 2 | 0 | 0 | 0 | 0

18. Primary Outcome: Urine Potential of Hydrogen (pH) Analysis by Dipstick Method for Part A
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by method up to 72 hours in Part A. Only those participants with data available at the indicated time points were analyzed.
Time Frame: Up to 72 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5
pH
  pH at Day -1 | 6.08 (0.469) | 6.00 (0.548) | 5.50 (0.548) | 5.92 (0.492) | 6.70 (1.483)
  pH at 24 hours | 6.04 (0.498) | 6.50 (0.447) | 5.83 (0.258) | 6.08 (0.204) | 6.80 (1.095)
  pH at 72 hours | 6.46 (0.753) | 6.00 (1.095) | 5.92 (0.492) | 6.42 (0.665) | 7.30 (0.671)

19. Primary Outcome: Number of Participants With Abnormal Urinalysis Parameters for Part B
Description: Urinalysis included dipstick urine test which was used to screen for glucose, ketones, occult blood and protein up to 14 days post dose The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose, ketones, occult blood and protein can be read as negative, trace, trace-intact, trace-lysed, 1+ and 2+ indicating proportional concentrations in the urine sample. Only categories with non-negative values have been presented. Only those participants available at the specified time points were analyzed represented by n=x in the category titles. Period 1 = Cohort 1 in Part B, Period 2 = Cohort 2 in Part B.
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
Participants
  Day -1, Ketones, Trace,n=2,7,0: number analyzed (Participants) | 2 | 7 | 0
  Day -1, Ketones, Trace,n=2,7,0 | 0 | 1 |
  Day -1, Occult blood,Trace-intact,n=2,7,0: number analyzed (Participants) | 2 | 7 | 0
  Day -1, Occult blood,Trace-intact,n=2,7,0 | 1 | 0 |
  Day 14, Ketones, Trace,n=2,7,0: number analyzed (Participants) | 2 | 7 | 0
  Day 14, Ketones, Trace,n=2,7,0 | 0 | 1 |
  Day 14, protein, 1+,n=2,7,0: number analyzed (Participants) | 2 | 7 | 0
  Day 14, protein, 1+,n=2,7,0 | 0 | 1 |
  Day -1,Occult blood,Trace-intact,n=2,0,8: number analyzed (Participants) | 2 | 0 | 8
  Day -1,Occult blood,Trace-intact,n=2,0,8 | 1 |  | 2
  Day 6,Occult blood,Trace-intact,n=2,0,8: number analyzed (Participants) | 2 | 0 | 8
  Day 6,Occult blood,Trace-intact,n=2,0,8 | 0 |  | 1
  Day 6,Occult blood,Trace-lysed,n=2,0,8: number analyzed (Participants) | 2 | 0 | 8
  Day 6,Occult blood,Trace-lysed,n=2,0,8 | 0 |  | 2
  Day 10, Ketones, Trace,n=2,0,8: number analyzed (Participants) | 2 | 0 | 8
  Day 10, Ketones, Trace,n=2,0,8 | 0 |  | 1
  Day 14, Protein, 2+,n=2,0,8: number analyzed (Participants) | 2 | 0 | 8
  Day 14, Protein, 2+,n=2,0,8 | 0 |  | 1
  Follow-up (week 8), Ketones, n=4,7,8 | 0 | 0 | 1
  Follow up (week 8), Occult blood, n=4,7,8 | 1 | 0 | 1
  Follow-up(week 8),Occult blood,Trace-lysed,n=4,7,8 | 0 | 0 | 2

20. Primary Outcome: Urine pH Analysis by Dipstick Method for Part B
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by method up to 8 weeks in Part B. Only those participants available at the specified time points were analyzed represented by n=x in the category titles. Period 1 = Cohort 1 in Part B, Period 2 = Cohort 2 in Part B.
Time Frame: Up to 8 weeks
Population: Safety Population for Part B
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part B-Matching Placebo | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 4 | 7 | 8
pH
  pH, Period 1, Day -1, n=2, 7, 0: number analyzed (Participants) | 2 | 7 | 0
  pH, Period 1, Day -1, n=2, 7, 0 | 6.25 (0.354) | 6.71 (0.906) |
  pH, Period 1, Day 4, n= 2, 7, 0: number analyzed (Participants) | 2 | 7 | 0
  pH, Period 1, Day 4, n= 2, 7, 0 | 6.25 (0.354) | 5.79 (0.393) |
  pH, Period 1, Day 6, n=2, 7, 0: number analyzed (Participants) | 2 | 7 | 0
  pH, Period 1, Day 6, n=2, 7, 0 | 6.25 (0.354) | 6.43 (0.535) |
  pH, Period 1, Day 10, n=2, 7, 0: number analyzed (Participants) | 2 | 7 | 0
  pH, Period 1, Day 10, n=2, 7, 0 | 6.25 (0.354) | 6.14 (0.244) |
  pH, Period 1, Day 14, n=2, 7, 0: number analyzed (Participants) | 2 | 7 | 0
  pH, Period 1, Day 14, n=2, 7, 0 | 6.75 (0.354) | 7.00 (0.957) |
  pH, Period 2, Day -1, n=2, 0, 8: number analyzed (Participants) | 2 | 0 | 8
  pH, Period 2, Day -1, n=2, 0, 8 | 6.50 (0.707) |  | 6.81 (0.594)
  pH, Period 2, Day 4, n=2, 0, 8: number analyzed (Participants) | 2 | 0 | 8
  pH, Period 2, Day 4, n=2, 0, 8 | 5.50 (0.707) |  | 6.25 (0.378)
  pH, Period 2, Day 6, n=2, 0, 8: number analyzed (Participants) | 2 | 0 | 8
  pH, Period 2, Day 6, n=2, 0, 8 | 6.50 (0.000) |  | 6.69 (0.458)
  pH, Period 2, Day 10, n=2, 0, 8: number analyzed (Participants) | 2 | 0 | 8
  pH, Period 2, Day 10, n=2, 0, 8 | 6.00 (0.000) |  | 6.38 (0.354)
  pH, Period 2, Day 14, n=2, 0, 8: number analyzed (Participants) | 2 | 0 | 8
  pH, Period 2, Day 14, n=2, 0, 8 | 6.00 (0.000) |  | 6.38 (0.582)
  pH, Follow-up (week 8), n=4, 7, 8 | 6.63 (0.750) | 6.29 (0.488) | 6.88 (0.744)

21. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-t]) Following Single Dose Administration of GSK3036656 for Part A
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 Ethylenediaminetetraacetic acid (EDTA) tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. The actual date and time of each blood sample collection was recorded. PK population comprised of participants in the Safety population who administered at least one dose of active treatment and had at least one evaluable PK sample.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hour*nanograms/milliliter | 771.0468 (26.0) | 3252.9152 (24.1) | 5686.4151 (11.4) | 782.7766 (18.1)

22. Primary Outcome: AUC From Time Zero Extrapolated to Infinite Time (AUC[0-infinity]) of GSK3036656 Following Single Dose Administration for Part A
Description: Cmax will be derived from the PK samples collected at the indicated time points Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. The actual date and time of each blood sample collection was recorded.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hour*nanograms/milliliter | 1404.5416 (29.9) | 3796.1488 (19.8) | 6557.7764 (13.8) | 1450.7468 (9.4)

23. Primary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) of GSK3036656 Following Single Dose Administration for Part A
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. The actual date and time of each blood sample collection was recorded.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanograms/milliliter | 49.06 (30.5) | 177.61 (23.1) | 207.38 (18.5) | 47.37 (23.5)

24. Primary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) of GSK3036656 Following Single Dose Administration for Part A
Description: as for outcome 23
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Median (Full Range); unit: hours
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours | 1.250 [0.50 to 1.50] | 1.000 [0.50 to 2.00] | 0.875 [0.75 to 2.00] | 2.000 [1.00 to 4.00]

25. Primary Outcome: Apparent Terminal Half-life (t1/2) of GSK3036656 Following Single Dose Administration for Part A
Description: as for outcome 23
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Median (Full Range); unit: hours
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours | 38.3230 [25.632 to 70.970] | 28.4128 [24.462 to 32.497] | 47.9680 [35.996 to 67.360] | 32.4248 [30.449 to 46.455]

26. Primary Outcome: AUC[0-t] Following Repeated Dose Administration of GSK3036656 for Part B
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1. The actual date and time of each blood sample collection was recorded. Results presented are for Day 1.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
hour*nanograms/milliliter | 485.5625 (12.3) | 1891.0416 (9.9)

27. Primary Outcome: AUC From Time Zero During a Dosing Interval of Duration Tau (AUC[0-tau]) of GSK3036656 Following Repeated Dose Administration for Part B
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14The actual date and time of each blood sample collection was recorded. Results presented are for Day 14.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
hour*nanograms/milliliter | 1392.2221 (12.5) | 4461.2565 (23.7)

28. Primary Outcome: Cmax of GSK3036656 Following Repeated Dose Administration for Part B
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1; at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14; and at pre-dose on Days 12 and 13. The actual date and time of each blood sample collection was recorded.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1; at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14; and at pre-dose on Days 12 and 13
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
nanograms/milliliter
  Day 1 | 48.40 (33.6) | 178.79 (32.8)
  Day 14 | 97.04 (19.8) | 309.55 (20.2)

29. Primary Outcome: Tmax of GSK3036656 Following Repeat Dose Administration for Part B
Description: as for outcome 28
Time Frame: as for outcome 28
Population: PK Population for Part B
Measure: Median (Full Range); unit: hours
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
hours
  Day 1 | 1.0000 [0.500 to 3.000] | 0.7500 [0.500 to 1.500]
  Day 14 | 0.7500 [0.500 to 1.500] | 0.7500 [0.500 to 1.500]

30. Primary Outcome: t1/2 of GSK3036656 Following Repeated Dose Administration for Part B
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14. The actual date and time of each blood sample collection was recorded. Results presented are for Day 14.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14.
Population: PK Population for Part B
Measure: Median (Full Range); unit: hours
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
hours | 40.1802 [30.843 to 66.636] | 34.5109 [24.758 to 54.625]

31. Secondary Outcome: AUC (0-t) of GSK3036656 Following Single Dose Administration in Fed Condition in Part A
Description: Blood samples for plasma PK analysis of GSK3036656 was collected into K3 EDTA tubes at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. The actual date and time of each blood sample collection was recorded. For the food effect assessment, the selected dose was given with a high fat meal.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours*nanograms/milliliter | 771.0468 (26.0) | 3252.9152 (24.1) | 5686.4151 (11.4) | 782.7766 (18.1)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 5 mg (Fed); Test type: Other; Ratio = 1.07, 90% CI 2-sided [0.87 to 1.34] — Mixed Effect Model has been used to assess Food Effect for the log transformed parameter AUC(0-t). Treatment in the fed/fasted state is fitted as Fixed Effect. Participant is fitted as Random Effect. Variance Components covariance structure is used

32. Secondary Outcome: AUC (0-infinity) of GSK3036656 Following Single Dose Administration in Fed Condition in Part A
Description: as for outcome 31
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours*nanograms/milliliter | 1404.5416 (29.9) | 3796.1488 (19.8) | 6557.7764 (13.8) | 1450.7468 (9.4)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 5 mg (Fed); Test type: Other; Ratio = 0.94, 90% CI 2-sided [0.71 to 1.26] — Mixed Effect Model has been used to assess Food Effect for the log transformed parameter AUC(0-inf). Treatment in the fed/fasted state is fitted as Fixed Effect. Participant is fitted as Random Effect. Variance Components covariance structure is use

33. Secondary Outcome: Cmax of GSK3036656 Following Single Dose Administration in Fed Condition in Part A
Description: as for outcome 31
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanograms/milliliter | 49.06 (30.5) | 177.61 (23.1) | 207.38 (18.5) | 35.54 (23.5)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 5 mg (Fed); Test type: Other; Ratio = 0.97, 90% CI 2-sided [0.76 to 1.23] — Mixed Effect Model has been used to assess Food Effect for the log transformed parameter Cmax. Treatment in the fed/fasted state is fitted as Fixed Effect. Participant is fitted as Random Effect. Variance Components covariance structure is used

34. Secondary Outcome: t1/2 of GSK3036656 Following Single Dose Administration in Fed Condition in Part A
Description: as for outcome 31
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Median (Full Range); unit: hours
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours | 38.3230 [25.632 to 70.970] | 28.4128 [24.462 to 32.497] | 47.9680 [35.996 to 67.360] | 32.4248 [30.449 to 46.455]
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 5 mg (Fed); Test type: Other; Ratio = 0.89, 90% CI 2-sided [0.64 to 1.23] — Fixed Effect Model has been used to assess Food Effect for the log transformed parameter t1/2 Treatment in the fed/fasted state is fitted as Fixed Effect

35. Secondary Outcome: Tmax of GSK3036656 Following Single Dose Administration in Fed Condition in Part A
Description: as for outcome 31
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Median (Full Range); unit: hours
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours | 1.250 [0.50 to 1.50] | 1.000 [0.50 to 2.00] | 0.875 [0.75 to 2.00] | 2.000 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 5 mg (Fed); Test type: Other; Median Difference (Final Values) = 0.75, 90% CI 2-sided [-0.50 to 2.50] — Hodges-Lehmann estimation is used to calculate the 90% confidence interval

36. Secondary Outcome: Observed Accumulation Ratio Based on AUC (AUC [Ro]) of GSK3036656 in Part B
Description: AUC Ro was calculated as Day 14 AUC(0-tau)/Day 1 AUC(0-t), where t and tau= 24 hours.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1; at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
Ratio of AUC | 2.8672 (9.1) | 2.3592 (21.6)

37. Secondary Outcome: Observed Accumulation Ratio Based on Cmax (RCmax) of GSK3036656 in Part B
Description: Rcmax was calculated as Day 14 Cmax/Day 1 Cmax. Statistics has been presented on geometric least square means.
Time Frame: as for outcome 36
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
Ratio of Cmax | 2.0052 (24.3) | 1.7313 (26.7)

38. Secondary Outcome: Steady State Ratio (Rss) of GSK3036656 in Part B
Description: Rss was calculated as Day 14 AUC (0-tau)/Day 1 AUC (0-inf). It was not possible to calculate AUC(0-inf) on Day 1 for the repeat dosing period, therefore it was not possible to calculate the (Rss).Na indicates data was not available.
Time Frame: as for outcome 36
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
Ratio of AUC | NA (NA) — It was not possible to calculate AUC(0-inf) on Day 1 for the repeat dosing period, therefore it was not possible to calculate the steady state ratio (Rss). | NA (NA) — It was not possible to calculate AUC(0-inf) on Day 1 for the repeat dosing period, therefore it was not possible to calculate the steady state ratio (Rss).

39. Secondary Outcome: Trough Plasma Concentrations at the End of the Dosing Interval (Ctau) of GSK3036656 Following Repeat Dose Administrations in Part B
Description: Blood samples for the analysis of Ctau were collected at Day 1 (24 hours), Day 12 (Pre-dose ), Day 13 (Pre-dose ), Day 14 (Pre-dose), Day 14 (24 hours). Ctau samples collected were used to assess attainment of steady state. Statistics has been presented on geometric least square means.
Time Frame: Day 1 (24 hours), Day 12 (Pre-dose ), Day 13 (Pre-dose ), Day 14 (Pre-dose), Day 14 (24 hours)
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
nanograms/milliliter
  Day 1, 24 hours | 14.32 (10.8) | 57.69 (10.5)
  Day 12, Pre-dose | 38.31 (20.8) | 139.14 (21.6)
  Day 13, Pre-dose | 41.78 (14.5) | 131.77 (28.8)
  Day 14, Pre-dose | 43.66 (15.1) | 139.54 (32.5)
  Day 14, 24 hours | 44.34 (14.8) | 139.25 (28.2)
Statistical Analysis 1: Comparison: Part B-Repeat GSK3036656 5 mg; Repeat GSK3036656 5mg Day 1-14; Test type: Other; Slope = 1.10, 90% CI 2-sided [1.09 to 1.10] — Mixed Effect Model has been used to assess Steady State. Day is fitted as a Fixed Effect. Participant is fitted as Random Effect Variance Components covariance structure is used
Statistical Analysis 2: Comparison: Part B-Repeat GSK3036656 15 mg; Repeat GSK3036656 15mg Day 1-14; Test type: Other; Slope = 1.08, 90% CI 2-sided [1.07 to 1.08] — [estimate comment as in outcome 39, analysis 1]

40. Secondary Outcome: AUC (0-infinity) as a Measure of Dose Proportionality of GSK3036656 Following Single Dose Administrations for Part A
Description: Blood samples for the analysis of AUC (0-infinity) were collected at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. AUC(0-infinity) following single doses was used for assessment of dose proportionality.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours*nanograms/milliliter | 1404.5416 (29.9) | 3796.1488 (19.8) | 6557.7764 (13.8) | 1450.7468 (9.4)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 15 mg; Test type: Other; Slope = 0.96, 90% CI 2-sided [0.82 to 1.10] — A slope of 1 indicates the pharmacokinetics are dose proportional. A slope greater than 1 indicates the increase in PK is greater than proportional to dose; Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect and Participant is fitted as Random Effect. An Unstructured covariance structure is used

41. Secondary Outcome: AUC (0-t) as a Measure of Dose Proportionality of GSK3036656 Following Single Dose Administrations for Part A
Description: Blood samples for the analysis of AUC (0-t) were collected at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. AUC(0-t) following single doses was used for assessment of dose proportionality.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours*nanograms/milliliter | 771.0468 (26.0) | 3252.9152 (24.1) | 5686.4151 (11.4) | 782.7766 (18.1)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 15 mg; Test type: Other; Slope = 1.32, 90% CI 2-sided [1.24 to 1.39] — Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect and Participant is fitted as Random Effect. An Unstructured covariance structure is used

42. Secondary Outcome: Cmax as a Measure of Dose Proportionality of GSK3036656 Following Single Dose Administrations for Part A
Description: Blood samples for the analysis of Cmax were collected at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1 in each period. Cmax following single doses was used for assessment of dose proportionality.
Time Frame: as for outcome 21
Population: PK Population for Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 5
hours*nanograms/milliliter | 49.06 (30.5) | 177.61 (23.1) | 207.38 (18.5) | 47.37 (23.5)
Statistical Analysis 1: Comparison: Part A-GSK3036656 5 mg vs Part A-GSK3036656 15 mg; Test type: Other; Slope = 0.96, 90% CI 2-sided [0.81 to 1.11] — [estimate comment as in outcome 41, analysis 1]

43. Secondary Outcome: AUC (0-tau) as a Measure of Dose Proportionality of GSK3036656 Following Repeat Dose Administrations for Part B
Description: Blood samples for the assessment of AUC (0-tau) were collected at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1; at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14; and at pre-dose on Days 12 and 13. AUC (0-tau) following repeat doses was used for assessment of dose proportionality.
Time Frame: as for outcome 28
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
hours*nanograms/milliliter | 1392.2221 (12.5) | 4461.2565 (23.7)
Statistical Analysis 1: Comparison: Part B-Repeat GSK3036656 5 mg vs Part B-Repeat GSK3036656 15 mg; Test type: Other; Slope = 1.24, 90% CI 2-sided [1.15 to 1.33] — Day 1.Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect
Statistical Analysis 2: Comparison: Part B-Repeat GSK3036656 5 mg vs Part B-Repeat GSK3036656 15 mg; Test type: Other; Slope = 1.06, 90% CI 2-sided [0.90 to 1.22] — Day 14. Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect

44. Secondary Outcome: Cmax as a Measure of Dose Proportionality of GSK3036656 Following Repeat Dose Administrations for Part B
Description: Blood samples for the assessment of Cmax were collected at Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 1; at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hour post-dose on Day 14; and at pre-dose on Days 12 and 13. Cmax following repeat doses was used for assessment of dose proportionality.
Time Frame: as for outcome 28
Population: PK Population for Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part B-Repeat GSK3036656 5 mg | Part B-Repeat GSK3036656 15 mg
Number analyzed (Participants) | 7 | 8
nanograms/milliliter
  Day 1 | 48.40 (33.6) | 178.79 (32.8)
  Day 14 | 97.04 (19.8) | 309.55 (20.2)
Statistical Analysis 1: Comparison: Part B-Repeat GSK3036656 5 mg vs Part B-Repeat GSK3036656 15 mg; Test type: Other; Slope = 1.19, 90% CI 2-sided [0.92 to 1.46] — Day 1. Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect
Statistical Analysis 2: Comparison: Part B-Repeat GSK3036656 5 mg vs Part B-Repeat GSK3036656 15 mg; Test type: Other; Slope = 1.06, 90% CI 2-sided [0.89 to 1.22] — Day 14. Power Model has been used to assess Dose Proportionality. Log-e(dose) is fitted as Fixed Effect

ADVERSE EVENTS:
Time Frame: nSAEs and SAEs were collected from Day -1 until 12 weeks in Part A and until 8 weeks in Part B.
Description: Safety Population was used to assess nSAEs and SAEs.
Groups:
- Part B-GSK3036656 5 mg: Participants received repeat dosing of GSK3036656 5 mg capsules orally once daily for 14 days.
- Part B-GSK3036656 15 mg: Participants received repeat dosing of GSK3036656 15 mg capsules orally once daily for 14 days.
Arm/Group | Part A-Matching Placebo | Part A-GSK3036656 5 mg | Part A-GSK3036656 15 mg | Part A-GSK3036656 25 mg | Part A-GSK3036656 5 mg (Fed) | Part B-Matching Placebo | Part B-GSK3036656 5 mg | Part B-GSK3036656 15 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/5 | 0/4 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/5 | 0/4 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 1/6 | 1/6 | 3/6 | 1/5 | 0/4 | 2/7 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-Matching Placebo (N=9) | Part A-GSK3036656 5 mg (N=6) | Part A-GSK3036656 15 mg (N=6) | Part A-GSK3036656 25 mg (N=6) | Part A-GSK3036656 5 mg (Fed) (N=5) | Part B-Matching Placebo (N=4) | Part B-GSK3036656 5 mg (N=7) | Part B-GSK3036656 15 mg (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03075410/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03075410/SAP_001.pdf